CLINICAL TRIAL: NCT03025386
Title: Establish a Concordance Between the Mismatch Negativity Amplitude and a Score of Logatoms Discrimination, Both Highlighting Capacities of Auditory Discrimination, in Adult Cochlear Implant Users
Brief Title: Establish a Concordance Between the Mismatch Negativity Amplitude and a Score of Logatoms Discrimination
Acronym: EVODA-ICMN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusions stopped
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL16_0196
Record Dates: First submitted 2017-01-16; First posted 2017-01-19 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2023-01

CONDITIONS: Cochlear Implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adult cochlear implant users (Other): Evaluation of a concordance between the mismatch negativity amplitude mesured by electroencephalography and the capacity of logatoms discrimination by using a logatoms test
  Interventions: Other: logatoms test; Other: Electroencephalography

INTERVENTIONS:
Other: logatoms test — A forced choice test will evaluate the discrimination of the most confusing logatoms in the cochlear implant users, and representative of the French language.
Other: Electroencephalography — Mesure of the mismatch negativity wave

SUMMARY:
A cochlear implant is a device for the rehabilitation of severe to profound hearing loss. Despite the standardization of surgical procedures and rehabilitation, speech discrimination performance varied significantly in cochlear implant users and could be improved by early individualized cares. However, there is no objective method yet to evaluate phonemes discrimination, especially in infants, which account for more than half of the indications for implantation. In electroencephalography (EEG), it is possible to highlight the discrimination of auditory stimuli studying the wave of MisMatch Negativity (MMN). In this work, this study propose to use the MMN as an objective vocal audiometry method to evaluate the ability to discriminate phonemes, the smallest units of oral language, in adult cochlear implant users.

DETAILED DESCRIPTION:
Context of the study Cochlear implant is an effective and recognized long-term solution for people with severe to profound neurosensory hearing loss. Its principle is to collect sounds of the environment, to analyze them, to transform them and, using an electrodes array placed in the cochlea, to transmit them back to the auditory nerve by electrical impulses. With practice, these are integrated and then recognized by the brain that associates a meaning. For normal hearing persons, speech recognition involves several time and frequency cues that the ear is able to decode. However, the cochlear implant distorts and alters some of these speech cues; the implant easily retransmits the temporal features but the frequency ones are much deteriorated. Thus, cochlear implant users preferentially use the temporal cues, which provide truncated and incomplete information, which often results in a lower quality understanding. Thus, learning or re-learning the language through the cochlear implant is difficult for the young deaf child as for the deaf adults.

The cochlear implant setting is essentially based on perceptual features. A detection threshold and a comfort level are fitting according to the perceptions of the patient and several objective tools. These provide important information but do not on the validity of the setting to ensure optimal speech understanding. The High Authority of Health suggests speech therapy in the overall rehabilitation of cochlear implant users. This aims to develop auditory skills according to four major perceptual axes: detection, identification, discrimination and understanding of sounds.

Despite these cares, cochlear implant users have speech recognition scores lower than those of normal-hearing people and have heterogeneous performances. Deafness etiology (auditory neuropathy, demyelization, ...), integrity of the auditory nerve, position of the electrode array in the cochlea, cognitive abilities, age implantation, duration of hearing loss, quality of cortical integration, cerebral plasticity, speech therapy, the family environment, implant fitting could affect subject performances.

Difficulties in speech understanding may be related to poor discrimination of phonemes, the smallest units of oral language. These phonemic confusions can be tested in adults by several tests such as the Phonetically Balanced Kindergarten test (PBK). However, in the very young child, childs with polyhandicap or the disabled adult, the evaluation of the language is more delicate and needs a long term.

Several electrophysiological techniques would nevertheless make it possible to objectively demonstrate the ability to discriminate phonemes in one measure. For example, the mismatch negativity wave (MMN) reflects a cognitive process showing the discrimination of two different sounds by the auditory system. It is measurable in adults and children, automatically and regardless of the level of vigilance. In this study use a MMN protocol to highlight phonemic discrimination capacities and then link them to subjective performances in the adult cochlear implant users. The first objective is to establish in these users a concordance between the amplitude of the MMN and a test of discrimination of logatoms, both highlighting the capacities of auditory discrimination. The second is to establish a concordance between the amplitude of the MMN and the scores obtained with the PBK.

Method

A forced choice test will evaluate the discrimination of the most confusing logatoms in the cochlear implant users, and representative of the French language. The following couples were selected:

* " fa " vs " sa "
* " la " vs " na "
* " pan " vs " pa "
* " pa " vs " ta "
* " pon " vs " po " Each couple of logatoms will be tested twenty times. If the score is greater than 16/20, the discrimination of logatoms pair will be considered positive. The test, carried out using Matlab MathWorks software, was automated so that the patient could do it without the intervention of the experimenter; It remains under its supervision in order to verify that the test is proceeding normally.

Obtaining the MMN requires a paradigm called "oddball", during which a "frequent" stimulus is emitted 80% of the time and a second stimulus called "deviant" is presented only 20% of the time. The high repetition rate of the frequent stimulus ("pa" for example) creates an electrophysiological baseline. When a deviant stimulus ("ba" for example) appears, this introduces a break in the electrophysiological baseline which results in the appearance of a so-called mismatch negative wave, the MMN. It shows the discrimination by the auditory system of two different stimuli. By studying the amplitude of this wave, it is possible to evaluate the quality of discrimination. A low or zero amplitude means that the subject did not discriminate the two logatoms. Conversely, the higher the amplitude, the greater the discrimination quality is. The wave latency can also be a variable to be observed. The earlier it is, the more it marks the ease of discrimination.

For each subject, the concordance with the score in the logatoms discrimination test will be analyzed separately for each pair. This will make it possible to evaluate the consistency of this concordance according to the pairs of tested logatoms. The optimal threshold of the MMN amplitude to identify subjects with good auditory discrimination is not yet known (innovative method). The first stage of our analysis will be to search for this threshold by constructing an receiver operating characteristic (ROC) curve to best distinguish patients with good and bad auditory discrimination in the test of the logatoms (choice of the threshold by the index of Youden). This threshold will then be used to classify subjects as having good or poor auditory discrimination according to the EEG. The agreement between the results of the EEG and the test of logatoms discrimination will then be analyzed by the calculation of a Kappa coefficient.

The PBK test will be used to evaluate an overall comprehension score. This test consists of 4 lists of 50 words respecting the occurrence of the phonemes of the French language and using mono- and bi-syllabic words. A score above 70% is accepted as a good performance. The concordance between the results of the EEG procedure for each logatoms (good and bad auditory discrimination defined as above) and the result of the PBK test will be analyzed using Kappa coefficients.

Finally, different secondary data will be collected: type of cochlear implant (mark, internal and external part), duration of implantation in months, etiology, data related to the implant setting (number of active electrodes , Thresholds C and T, IDR, automatic functions like SCAN, ADRO, ...)

ELIGIBILITY:
Inclusion criteria:

* Aged from 18 to 75
* Severe to profound deafness
* Cochlear implant user for over a year
* Affiliation or beneficiary of the social insurance

Exclusion criteria:

* Phonetically balanced kindergarten score less than 25%
* No steady setting
* Contralateral hearing aid
* Electroacoustic stimulation device or bilateral cochlear implant user
* Inactive electrodes > 3
* Cochlear Implant wore less than 7 hours per day
* Disorders of memory, attention or executive functions
* Associated disorders with deafness
* No informed consent
* Patient participating in other biomedical research
* Patient who has undergone cochlear reimplantation or brain surgery
* Withdrawal of consents
* Patient lost to follow-up
* Death

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Correlation between MMN amplitude and logatoms discrimination score in the discrimination capacity | 30 days
  The discrimination capacity (positive/ negative) defined by an MMN amplitude above a threshold will be estimated using a ROC curve based on the logatoms discrimination scores The discrimination capacity defined by logatoms test will be positive if the discrimination score is higher or equal to 80%.

SECONDARY OUTCOMES:
Correlation between MMN amplitude and the Phonetically Balanced Kindergarten score and Vocoder test | within the first 30 days after the first visit
  The discrimination capacity will be positive if the correlation score is higher or equal to 70%.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric VENAIL, PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No